CLINICAL TRIAL: NCT05422768
Title: PTSD Clinical Team Research Clinic (PCT Research Clinic)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB_00136053
Record Dates: First submitted 2022-02-16; First posted 2022-06-16 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: PTSD
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Warrior Renew: Warrior Renew is a program for military sexual trauma (MST).
  Interventions: Behavioral: Warrior Renew
- Warrior Renew + EAL: Warrior Renew and EAL are combined into one program for military sexual trauma (MST).
  Interventions: Behavioral: Warrior Renew + EAL

INTERVENTIONS:
Behavioral: Warrior Renew — Warrior Renew is a program for military sexual trauma (MST).
  Groups: Warrior Renew
Behavioral: Warrior Renew + EAL — Warrior Renew and EAL are combined into one program for military sexual trauma (MST).
  Groups: Warrior Renew + EAL

SUMMARY:
Part of the IRB_00136053 study was to look at the effectiveness of Warrior Renew and Warrior Renew+EAL interventions. Furthermore, demographic information on Veteran participants will be analyzed.

DETAILED DESCRIPTION:
EAL is one of a group of equine-assisted services (EAS), which are aimed at providing benefits for humans, including addressing emotional, mental and social components of functioning. In recent years, the use of EAS has grown rapidly in Europe and the United States in general and is being increasingly used for active-duty military and veteran Veteran populations. As we have previously reviewed, there is evidence that EAS, such as EAL, can contribute to reduction of PTSD and other psychological symptoms as well as enhancing well-being via improvements in resilience, life satisfaction, trust, self-image, and self-control, as well as quality of life.

ELIGIBILITY:
Inclusion Criteria:

* referred to PTSD team

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Veterans who were referred to PTSD team were contacted to see if they wanted to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-05-11 (Estimated); Study Completion 2024-05-11 (Estimated)

PRIMARY OUTCOMES:
Change in PCL Measures Pre to Post-Intervention and by Intervention Type | through study completion, an average of 2 years
  The Posttraumatic Checklist-5 (PCL) was used to assess self-reported symptoms of PTSD using items consistent with the Diagnostic and Statistical Manual - Fifth Edition. PCL-5 scores can range from 0 to 80 with higher score indicating more PTSD symptoms.
Change in PHQ Measures Pre to Post-Intervention and by Intervention Type | through study completion, an average of 2 years
  The Patient Health Questionnaire (PHQ) was used to assess symptoms of major depression. PHQ scores range from 0 to 27 with higher scores indicating greater depression symptoms.
Change in PTCI Measures Pre to Post-Intervention and by Intervention Type | through study completion, an average of 2 years
  The Posttraumatic Cognitions Inventory (PTCI) was used to assess trauma-related thoughts and beliefs. PTCI can range from 33-252 with higher scores indicating more distress.
Mean and Standard Deviation of Demographic information by Intervention Type | through study completion, an average of 2 years
  The demographic information analyzed includes age, sex, race, ethnicity, religion, service era, service connection, service connection percentage, diagnoses, Emergency Department (ED) visits, Inpatient Psychiatric Unit (IPU) visits, Substance Abuse Residential Rehabilitation Treatment Program (SARRTP) visits.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Roberge, PhD, Principal Investigator — Salt Lake City Veterans' Administration Medical Center
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, Utah, United States

REFERENCES:
- [Result] U.S. Congress. House Report 114-102: National Defense Authorization Act for Fiscal Year 2016; 2015. https://www.congress.gov/congressional-report/114th-congress/house-report/102/1
- [Result] Bachi K, Terkel J, Teichman M. Equine-facilitated psychotherapy for at-risk adolescents: the influence on self-image, self-control and trust. Clin Child Psychol Psychiatry. 2012 Apr;17(2):298-312. doi: 10.1177/1359104511404177. Epub 2011 Jul 14. PMID 21757481
- [Result] Ferruolo DM. Psychosocial Equine Program for Veterans. Soc Work. 2016 Jan;61(1):53-60. doi: 10.1093/sw/swv054. PMID 26897999
- [Result] Arnon S, Fisher PW, Pickover A, Lowell A, Turner JB, Hilburn A, Jacob-McVey J, Malajian BE, Farber DG, Hamilton JF, Hamilton A, Markowitz JC, Neria Y. Equine-Assisted Therapy for Veterans with PTSD: Manual Development and Preliminary Findings. Mil Med. 2020 Jun 8;185(5-6):e557-e564. doi: 10.1093/milmed/usz444. PMID 32034416
- [Result] Marchand WR, Andersen SJ, Smith JE, Hoopes KH, Carlson JK. Equine-Assisted Activities and Therapies for Veterans With Posttraumatic Stress Disorder: Current State, Challenges and Future Directions. Chronic Stress (Thousand Oaks). 2021 Feb 15;5:2470547021991556. doi: 10.1177/2470547021991556. eCollection 2021 Jan-Dec. PMID 33644617
- [Result] Shelef A, Brafman D, Rosing T, Weizman A, Stryjer R, Barak Y. Equine Assisted Therapy for Patients with Post Traumatic Stress Disorder: A Case Series Study. Mil Med. 2019 Oct 1;184(9-10):394-399. doi: 10.1093/milmed/usz036. PMID 30839068
- [Result] Burton LE, Qeadan F, Burge MR. Efficacy of equine-assisted psychotherapy in veterans with posttraumatic stress disorder. J Integr Med. 2019 Jan;17(1):14-19. doi: 10.1016/j.joim.2018.11.001. Epub 2018 Nov 16. PMID 30497951
- [Result] Malinowski K, Yee C, Tevlin JM, Birks EK, Durando MM, Pournajafi-Nazarloo H, Cavaiola AA, McKeever KH. The Effects of Equine Assisted Therapy on Plasma Cortisol and Oxytocin Concentrations and Heart Rate Variability in Horses and Measures of Symptoms of Post-Traumatic Stress Disorder in Veterans. J Equine Vet Sci. 2018 May;64:17-26. doi: 10.1016/j.jevs.2018.01.011. Epub 2018 Feb 12. PMID 30973147
- [Result] Johnson RA, Albright DL, Marzolf JR, Bibbo JL, Yaglom HD, Crowder SM, Carlisle GK, Willard A, Russell CL, Grindler K, Osterlind S, Wassman M, Harms N. Effects of therapeutic horseback riding on post-traumatic stress disorder in military veterans. Mil Med Res. 2018 Jan 19;5(1):3. doi: 10.1186/s40779-018-0149-6. PMID 29502529
- [Result] Steele E, Wood DS, J Usadi E, Applegarth DM. TRR's Warrior Camp: An Intensive Treatment Program for Combat Trauma in Active Military and Veterans of All Eras. Mil Med. 2018 Mar 1;183(suppl_1):403-407. doi: 10.1093/milmed/usx153. PMID 29635563
- [Result] Duncan CR, Critchley S, & Marland J. Can Praxis: A model of equine assisted learning (EAL) for PTSD. Canadian Military Journal. 2014; 14(2):64-69.
- [Result] Lanning BA, Krenek N. Guest Editorial: Examining effects of equine-assisted activities to help combat veterans improve quality of life. J Rehabil Res Dev. 2013;50(8):vii-xiii. doi: 10.1682/JRRD.2013.07.0159. No abstract available. PMID 24458903
- [Result] Lanning BA, Wilson AL, Krenek N, & Beaujean AA. Using therapeutic riding as an intervention for combat Veterans: An international classification of functioning, disability, and health (ICF) approach. Occupational Therapy in Mental Health. 2017; 33(3):259-278. https://doi.org/10.1080/0164212X.2017.1283282
- [Result] Sylvia L, West E, Blackburn AM, Gupta C, Bui E, Mahoney T, Duncan G, Wright EC, Lejeune S, Spencer TJ. Acceptability of an adjunct equine-assisted activities and therapies program for veterans with posttraumatic stress disorder and/or traumatic brain injury. J Integr Med. 2020 Mar;18(2):169-173. doi: 10.1016/j.joim.2020.01.005. Epub 2020 Jan 21. PMID 31996299
- [Result] Wharton T, Whitworth J, Macauley E, Malone M. Pilot testing a manualized equine-facilitated cognitive processing therapy (EF-CPT) intervention for PTSD in veterans. Psychiatr Rehabil J. 2019 Sep;42(3):268-276. doi: 10.1037/prj0000359. Epub 2019 Mar 25. PMID 30907609
- [Result] Cerulli C, Minganti C, De Santis C, Tranchita E, Quaranta F, Parisi A. Therapeutic horseback riding in breast cancer survivors: a pilot study. J Altern Complement Med. 2014 Aug;20(8):623-9. doi: 10.1089/acm.2014.0061. Epub 2014 Jun 25. PMID 24963599
- [Result] Fields B, Bruemmer J, Gloeckner G, Wood W. Influence of an Equine-Assisted Activities Program on Dementia-Specific Quality of Life. Am J Alzheimers Dis Other Demen. 2018 Aug;33(5):309-317. doi: 10.1177/1533317518772052. Epub 2018 May 9. PMID 29742908